CLINICAL TRIAL: NCT07074860
Title: Clinical Screening and Peer Interventions to Prevent Substance Use in At-Risk Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Constance van Eeghen, Associate Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003562; AWD00001448 (Other Grant/Funding Number: NIDA Challenge Grant Award)
Record Dates: First submitted 2025-07-01; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Initation of Substance Use Disorder
Keywords: Substance use prevention; Peer to peer support for adolescents; Video-based awareness raising

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer to peer video (Experimental): This study involves the pilot testing of novel substance use prevention videos, which are in the process of being developed for this study by a local group of adolescents that have created teen-focused public health messaging.
  Interventions: Behavioral: Peer to peer video to raise awareness about substance use

INTERVENTIONS:
Behavioral: Peer to peer video to raise awareness about substance use — A total of 4 short, animated videos will be created using design concepts and language created by the VT RAYS. Each video will be <2 minutes in length and address a specific topic including e-cigarette, cannabis, alcohol and other substance use. These videos will be curated online and shown to study participants during their scheduled primary care visits. The video will be followed by a short online survey available immediately after viewing to collect feedback on the content.

SUMMARY:
The goal of this clinical trial is to test a method of preventing substance use among adolescents. Young people aged 11-14 who have depression, anxiety, or attention deficit hyperactivity disorder (ADHD) are at higher than usual risk for starting substances such as alcohol, tobacco products, or drugs. The main question the investigators aim to answer is:

"Will watching short videos in their doctor's office every three months that were made by other adolescents in their community about not using drugs and other substances prevent at risk adolescents from starting to use those substances?"

The investigators will measure the outcome by asking participants to complete a survey every three months. The survey is a standard set of questions about behavior, including substance use. If they have started to use substances, they will get treatment for substance use. If they have not, they will watch another video and come back three months later to repeat the survey.

DETAILED DESCRIPTION:
Adolescent substance use is a significant public health concern with self-reported use of drugs and/or alcohol remaining high in the United States. Data from the National Survey on Drug Use and Health show that adolescent initiation of alcohol and cannabis use in the past year was 9.1% and 5.4% respectively. Evidence suggests that earlier initiation of substance use is linked to higher rates of substance use disorder (SUD) in adulthood. The American Academy of Pediatrics (AAP) recommends substance use screening for adolescents beginning at age 11 at annual health supervision visits. The Substance Abuse and Mental Health Services Administration (SAMHSA) also provides recommendations on screening for adolescent substance use using validated screening tools. Validated tools for adolescent substance use screening are available to primary care providers (PCPs) to administer to patients at health supervision visits. To use these resources effectively, practices are encouraged to have a pathway for administering screening tools and addressing responses. The screening, brief intervention, and referral to treatment (SBIRT) model is recommended as the ideal clinician response to positive screening. Negative screens for substance use generally are addressed with motivational interviewing but might not be discussed during a busy health supervision visit if there are other concerns to address. Furthermore, PCP delivered brief interventions have been shown to have mixed results providing some benefit in decreasing heavy alcohol use, but not cannabis use or abstinence.

Several common mental health diagnoses are associated with increased risk of adolescent substance use including depression, anxiety, and attention deficit hyperactivity disorder (ADHD). Adolescents receiving treatment for these diagnoses from their PCP often have frequent office visits ranging from monthly to quarterly. Screening and assessment tools are often utilized to both diagnose and monitor response to treatment for these conditions. Commonly used tools include the Patient Health Questionnaire 9 (PHQ-9) modified for teens for depression, Generalized Anxiety Disorder 7 (GAD-7) for anxiety, and NICHQ Vanderbilt scales for ADHD. Currently, there are no recommendations to screen more frequently for substance use in adolescents with depression, anxiety and/or ADHD despite their increased risk of developing SUD.

Recent Interventions: Many interventions for adolescent substance use prevention have been developed and studied. A recent study found that computer-based screening of adolescents for alcohol and cannabis followed by a brief educational intervention decreased risk behaviors in those reporting current use, but no benefit in those reporting no use. This study provided adolescents with immediate calculation of their reported use followed by multiple pages of scientific data and vignettes, focusing on decreasing risky use and riding with an impaired driver. However, a recent meta-analysis of primary prevention programs including Life Skills Training and other models, have demonstrated variable results and benefits. Similarly, meta-analysis of school-based interventions for alcohol and cannabis use in adolescents provided low or very-low quality evidence of effectiveness. Brief interventions targeting adolescents with depression and anxiety have not shown clear benefits in decreasing substance use, in part due to variability of models and interventions evaluated. Each of these studies concluded more research was needed to determine effectiveness of individual models in decreasing risk behaviors or preventing substance use.

Peer-based interventions have shown utility for improving adolescent engagement and participation in their health care, including the Providers and Teens Communicating for Health (PATCH) program. Studies of similar programs provide supporting evidence. One study examined a peer support service for youth experiencing complex challenges with mental health, physical health and/or substance use to better understand key features and underlying mechanisms that lead to improved client outcomes, noting the importance of mechanisms related to 1) positive identity development through identification with peers, 2) enhanced social connections, 3) observational learning and 4) enhanced autonomy and empowerment. Another looked at the direct relation between positive peer affiliation and substance use, and whether positive peer affiliation moderated the relation between self-reported sensation-seeking, future orientation, self-regulation and substance use, finding that having friends who generally engage in positive activities is an important buffer against socioemotional risk factors. Building on previous research, another examined the relationship of positive peer influence with indices of substance use and compared abstinent adolescents and substance-using adolescents on positive peer influence, with the results identifying positive peer influence as a significant predictor of lower substance use behaviors in adolescents and with positive influence from close friends being the strongest predictor. These findings, while hopeful, have been shown to need more study in sub-group analysis, as results vary by gender and other characteristics.

Looking more specifically at studies that examine the impact of peer-based interventions on prevention of substance use in adolescents, a systematic review of the literature on prevention of substance initiation for ages 11-21 showed peer-led interventions were associated with benefit in relation to alcohol use (OR = 0.80, 95% CI = 0.65-0.99, P = 0.036), while three studies ( n = 976 students in 38 schools) suggested an association with lower odds of cannabis use (OR = 0.70, 0.50-0.97, P = 0.034)17. Additional studies confirmed the value of this approach, with sometimes mixed results in sub-group analysis.

Proposed Model: Clinical Screening and Peer Interventions to Prevent Substance Use in At-Risk Adolescents: The investigators propose trialing an intervention focused on prevention of substance use among adolescents aged 11-14 at increased risk due to depression, anxiety, or ADHD diagnoses and who have not initiated substance use. These at-risk patients are routinely scheduled for regular follow-up visits with their PCPs for management of their mental health diagnoses. With our model, they will be rescreened for substance use quarterly (rather than annually) to promote more frequent conversations about prevention with their providers. They will receive access to brief video modules about avoiding substance use made by local peers.

This model is based on the novel use of clinical screening to identify at-risk adolescents not using substances for peer-led interactions. The use of video modules for substance use prevention is well-supported in the literature, as are social media awareness campaigns and media literacy for adolescents. Recently, the American Psychological Association issued recommendations for skill training for adolescents "to ensure that youth have skills that will maximize the chances for balanced, safe and meaningful experiences" using social media. The proposed intervention provides more frequent screening for substance use initiation to promote more frequent conversations about prevention with their providers and access to brief video modules about avoiding substance use made by local peers.

The primary objective of this study is to develop and trial an intervention of peer-designed and peer-delivered videos focused on prevention of substance use for adolescents aged 11-14 who have diagnosed depression, anxiety, or ADHD and who have not initiated substance use.

The secondary objective is to obtain user feedback on the videos for later development in a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depression, anxiety, or ADHD

Exclusion Criteria:

* Has not initiated substance use

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
CRAFFT 2.1 Questionnaire total score | Up to 12 months after enrollment
  The CRAFFT 2.1 questionnaire is a substance use screening tool for pediatric patients age 11 and older. It is recommended by the US Preventative Services Task Force and American Academy of Pediatrics and has been validated for use in adolescents.

SECONDARY OUTCOMES:
Video Feedback Survey | Up to 12 months after enrollment
  4 items scored on a Likert Scale (Strongly disagree to Strongly agree) assessing whether the video provided new information, was interesting, was recommended for others of the same age, and whether the participant felt comfortable talking to their healthcare provider about using alcohol and drugs.

IPD SHARING:
Plan to Share IPD: No
This is a pilot study for proof of concept. The tertiary purpose of the study is to support a larger test of the intervention, if found beneficial.

REFERENCES:
- [Background] Winn LAP, Paquette KL, Donegan LRW, Wilkey CM, Ferreira KN. Enhancing adolescent SBIRT with a peer-delivered intervention: An implementation study. J Subst Abuse Treat. 2019 Aug;103:14-22. doi: 10.1016/j.jsat.2019.05.009. Epub 2019 May 14. PMID 31229188
- [Background] Giambra, D.M., Adolescent peer support groups to reduce risky behaviors. Dissertation Abstracts International: Section B: The Sciences and Engineering. Vol. 83(5B). 2022
- [Background] Mitchell SG, Kelly SM, Gryczynski J, Myers CP, O'Grady KE, Kirk AS, Schwartz RP. The CRAFFT cut-points and DSM-5 criteria for alcohol and other drugs: a reevaluation and reexamination. Subst Abus. 2014;35(4):376-80. doi: 10.1080/08897077.2014.936992. PMID 25036144
- [Background] Knight JR, Sherritt L, Shrier LA, Harris SK, Chang G. Validity of the CRAFFT substance abuse screening test among adolescent clinic patients. Arch Pediatr Adolesc Med. 2002 Jun;156(6):607-14. doi: 10.1001/archpedi.156.6.607. PMID 12038895
- [Background] Greene K, Ray AE, Choi HJ, Glenn SD, Lyons RE, Hecht ML. Short term effects of the REAL media e-learning media literacy substance prevention curriculum: An RCT of adolescents disseminated through a community organization. Drug Alcohol Depend. 2020 Sep 1;214:108170. doi: 10.1016/j.drugalcdep.2020.108170. Epub 2020 Jul 10. PMID 32693198
- [Background] Kupersmidt JB, Scull TM, Benson JW. Improving media message interpretation processing skills to promote healthy decision making about substance use: the effects of the middle school media ready curriculum. J Health Commun. 2012;17(5):546-63. doi: 10.1080/10810730.2011.635769. Epub 2012 Feb 16. PMID 22339322
- [Background] Park E, Jang BG. Youth Substance Use Prevention Using Disciplinary Literacy Strategies: A Pilot Study. J Addict Nurs. 2018 Oct/Dec;29(4):235-243. doi: 10.1097/JAN.0000000000000253. PMID 30507819
- [Background] Wang, T.-C., F.-C. Chang, C.-H. Lee, H.-Y. Chi, L.-J. Huang, and C.-C. Tseng, Adolescents' misperceptions and low literacy associated with the inappropriate use of over-the-counter cold medicines. Journal of Substance Use, 2020. 25(1): p. 101-106
- [Background] Kaestle CE, Chen Y, Estabrooks PA, Zoellner J, Bigby B. Pilot evaluation of a media literacy program for tobacco prevention targeting early adolescents shows mixed results. Am J Health Promot. 2013 Jul-Aug;27(6):366-9. doi: 10.4278/ajhp.120221-ARB-105. Epub 2013 Mar 4. PMID 23458374
- [Background] Primack BA, Douglas EL, Land SR, Miller E, Fine MJ. Comparison of media literacy and usual education to prevent tobacco use: a cluster-randomized trial. J Sch Health. 2014 Feb;84(2):106-15. doi: 10.1111/josh.12130. PMID 25099425
- [Background] Shensa A, Phelps-Tschang J, Miller E, Primack BA. A randomized crossover study of web-based media literacy to prevent smoking. Health Educ Res. 2016 Feb;31(1):48-59. doi: 10.1093/her/cyv062. Epub 2015 Dec 16. PMID 26675176
- [Background] Bier MC, Zwarun L, Sherblom SA. Evidence of the Value of the Smoking Media Literacy Framework for Middle School Students. J Sch Health. 2016 Oct;86(10):717-25. doi: 10.1111/josh.12425. PMID 27619762
- [Background] Bonar EE, Bauermeister JA, Blow FC, Bohnert ASB, Bourque C, Coughlin LN, Davis AK, Florimbio AR, Goldstick JE, Wisnieski DM, Young SD, Walton MA. A randomized controlled trial of social media interventions for risky drinking among adolescents and emerging adults. Drug Alcohol Depend. 2022 Aug 1;237:109532. doi: 10.1016/j.drugalcdep.2022.109532. Epub 2022 Jun 11. PMID 35759874
- [Background] Bonyani A, Safaeian L, Chehrazi M, Etedali A, Zaghian M, Mashhadian F. A high school-based education concerning drug abuse prevention. J Educ Health Promot. 2018 Jul 6;7:88. doi: 10.4103/jehp.jehp_122_17. eCollection 2018. PMID 30079359
- [Background] Hopson L, Wodarski J, Tang N. The effectiveness of electronic approaches to substance abuse prevention for adolescents. J Evid Inf Soc Work. 2015;12(3):310-22. doi: 10.1080/15433714.2013.857178. Epub 2015 Jan 28. PMID 25661894
- [Background] Shin Y, Miller-Day M, Hecht ML, Krieger JL. Entertainment-Education Videos as a Persuasive Tool in the Substance Use Prevention Intervention "keepin' it REAL". Health Commun. 2018 Jul;33(7):896-906. doi: 10.1080/10410236.2017.1321163. Epub 2017 Jun 6. PMID 28586239
- [Background] Abraham O, Szela L, Brasel K, Hoernke M. Engaging youth in the design of prescription opioid safety education for schools. J Am Pharm Assoc (2003). 2022 Mar-Apr;62(2):441-449. doi: 10.1016/j.japh.2021.10.016. Epub 2021 Oct 20. PMID 34736864
- [Background] Dobbie F, Purves R, McKell J, Dougall N, Campbell R, White J, Amos A, Moore L, Bauld L. Implementation of a peer-led school based smoking prevention programme: a mixed methods process evaluation. BMC Public Health. 2019 Jun 13;19(1):742. doi: 10.1186/s12889-019-7112-7. PMID 31196124
- [Background] Demirezen, D., A. Karaca, D. Konuk Sener, and H. Ankarali, Agents of Change: The Role of the Peer Education Program in Preventing Adolescent Substance Abuse. Journal of Child & Adolescent Substance Abuse, 2019. 28(5): p. 376-387
- [Background] Golonka MM, Peairs KF, Malone PS, Grimes CL, Costanzo PR. Natural Peer Leaders as Substance Use Prevention Agents: the Teens' Life Choice Project. Prev Sci. 2017 Jul;18(5):555-566. doi: 10.1007/s11121-017-0790-4. PMID 28500558
- [Background] Georgie J M, Sean H, Deborah M C, Matthew H, Rona C. Peer-led interventions to prevent tobacco, alcohol and/or drug use among young people aged 11-21 years: a systematic review and meta-analysis. Addiction. 2016 Mar;111(3):391-407. doi: 10.1111/add.13224. PMID 26518976
- [Background] Kwan PP, Sussman S, Valente TW. Peer leaders and substance use among high-risk adolescents. Subst Use Misuse. 2015 Feb;50(3):283-91. doi: 10.3109/10826084.2014.977395. Epub 2014 Nov 19. PMID 25407377
- [Background] Beard SJ, Wolff JM. The moderating role of positive peers in reducing substance use in college students. J Am Coll Health. 2022 May-Jun;70(4):1059-1070. doi: 10.1080/07448481.2020.1784907. Epub 2020 Jul 16. PMID 32669053
- [Background] Halsall T, Daley M, Hawke L, Henderson J, Matheson K. "You can kind of just feel the power behind what someone's saying": a participatory-realist evaluation of peer support for young people coping with complex mental health and substance use challenges. BMC Health Serv Res. 2022 Nov 16;22(1):1358. doi: 10.1186/s12913-022-08743-3. PMID 36384511
- [Background] McDanal R, Parisi D, Opara I, Schleider JL. Effects of Brief Interventions on Internalizing Symptoms and Substance Use in Youth: A Systematic Review. Clin Child Fam Psychol Rev. 2022 Jun;25(2):339-355. doi: 10.1007/s10567-021-00372-2. Epub 2021 Nov 3. PMID 34731373
- [Background] Carney T, Myers BJ, Louw J, Okwundu CI. Brief school-based interventions and behavioural outcomes for substance-using adolescents. Cochrane Database Syst Rev. 2016 Jan 20;2016(1):CD008969. doi: 10.1002/14651858.CD008969.pub3. PMID 26787125
- [Background] Tremblay M, Baydala L, Khan M, Currie C, Morley K, Burkholder C, Davidson R, Stillar A. Primary Substance Use Prevention Programs for Children and Youth: A Systematic Review. Pediatrics. 2020 Sep;146(3):e20192747. doi: 10.1542/peds.2019-2747. Epub 2020 Aug 7. PMID 32769198
- [Background] Knight JR, Sherritt L, Gibson EB, Levinson JA, Grubb LK, Samuels RC, Silva T, Vernacchio L, Wornham W, Harris SK. Effect of Computer-Based Substance Use Screening and Brief Behavioral Counseling vs Usual Care for Youths in Pediatric Primary Care: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2019 Jun 5;2(6):e196258. doi: 10.1001/jamanetworkopen.2019.6258. PMID 31225897
- [Background] Klein RJ, Gyorda JA, Jacobson NC. Anxiety, depression, and substance experimentation in childhood. PLoS One. 2022 May 24;17(5):e0265239. doi: 10.1371/journal.pone.0265239. eCollection 2022. PMID 35609016
- [Background] Steele DW, Becker SJ, Danko KJ, Balk EM, Adam GP, Saldanha IJ, Trikalinos TA. Brief Behavioral Interventions for Substance Use in Adolescents: A Meta-analysis. Pediatrics. 2020 Oct;146(4):e20200351. doi: 10.1542/peds.2020-0351. Epub 2020 Sep 14. PMID 32928988
- [Background] Levy SJ, Williams JF; COMMITTEE ON SUBSTANCE USE AND PREVENTION. Substance Use Screening, Brief Intervention, and Referral to Treatment. Pediatrics. 2016 Jul;138(1):e20161211. doi: 10.1542/peds.2016-1211. Epub 2016 Jun 20. PMID 27325634
- [Background] Bright Futures: Guidelines for Health Supervision of Infants, Children and Adolescents. 4th ed. 2017: American Academy of Pediatrics
- [Background] Groenman AP, Janssen TWP, Oosterlaan J. Childhood Psychiatric Disorders as Risk Factor for Subsequent Substance Abuse: A Meta-Analysis. J Am Acad Child Adolesc Psychiatry. 2017 Jul;56(7):556-569. doi: 10.1016/j.jaac.2017.05.004. Epub 2017 May 11. PMID 28647007
- [Background] Center for Behavioral Health Statistics and Quality, S.A.a.M.H.S.A., Behavioral health equity report 2021: Substance use and mental health indicators measured from the National Survey on Drug Use and Health (NSDUH), 2015-2019. 2021, Substance Abuse and Mental Health Services Administration: Rockville, MD.
- See also: McCabe, M.A. APA panel issues recommendations for adolescent social media use 2023 — https://www.apa.org/news/press/releases/2023/05/adolescent-social-media-use-recommendations